CLINICAL TRIAL: NCT05342285
Title: Flow Mediated Dilation in Association With Hyperuricemia as Predictors of Cardiovascular Affection in Patients With Systemic Lupus
Brief Title: Flow Mediated Dilation in Association With Hyperuricemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lobna Ahmed Hassan, principle investigator, Assiut University
Other Study IDs: FMD
Record Dates: First submitted 2022-03-21; First posted 2022-04-22 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: SLE; Cardiovascular Diseases; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- normal FMD: SLE femals patientd with normal flow mediated whose ages from 18 to 45yrs
  Interventions: Diagnostic Test: Flow mediated dilation
- abnormal FMD: SLE femals with abnormal flow mediated dikation ages between 18 to 45yrs old
  Interventions: Diagnostic Test: Flow mediated dilation
- Normal female: normal femals whise ages from 18 to 45yrs old
  Interventions: Diagnostic Test: Flow mediated dilation

INTERVENTIONS:
Diagnostic Test: Flow mediated dilation — flow mediated dilation in brachial artery

SUMMARY:
Assess cardiovascular affection and subclinical atherosclerosis in patients with systemic lupus using the non invasive flow mediated dilation.

evaluate the role of uric acid as independent marker of cardiovascular risk in systemic lupus patient

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a complex autoimmune disease that is characterized by multiple end-organ damage and predominantly affects premenopausal women.

Cardiovascular disease is a major cause of morbidity and mortality in systemic lupus erythematosus (SLE) patients. These patients have a higher incidence and an earlier age of onset of ischemic heart disease, carotid atherosclerosis, cerebrovascular stroke, and peripheral vascular Disease. Traditional cardiovascular risk factors, including hypertension, diabetes mellitus, dyslipidemia, and physical inactivity, only account partially for the elevated vascular risk in SLE patients .

Vascular stiffness proven to have better predictive value for fatal and non-fatal cardiovascular events than traditional risk factors in hypertensives and patients with end-stage renal disease or coronary artery disease . Endothelial dysfunction represents the initial step of atherosclerosis and correlates with arterial stiffness which is associated with incident cardiovascular events.

Brachial artery reactivity testing (BART) is used to noninvasively assess responsiveness to reactive hyperemia (flow-mediated dilation [FMD]) and evaluate nitric oxide [NO]-dependent large vessel endothelial function. Reduced FMD reflects impaired endothelial-dependent vasodilation indicative of vascular dysfunction.

Uric acid (UA), the final product of purine degradation, is formed in the liver from precursor proteins and is excreted by the kidneys and intestines. At physiologic concentrations, UA exhibits excellent antioxidant activity; however, when UA exceeds its physiologic levels, it can propagate oxidative damage. Furthermore, chronic elevation of UA constitutes a risk factor for many diseases, as it can promote inflammation and endothelial dysfunction .

Higher prevalence of hyperuricemia in patients with SLE might be owing to several endogenous and exogenous mechanisms such as inflammation, hypertension, and renal involvement, which are prevalent in patients with SLE and have been identified as provoking hyperuricemia through different mechanisms. On the contrary, increased levels of UA can aggravate inflammation, hypertension, and renal disease, thus creating a vicious cycle. Hyperactivity of the xanthine oxidase enzyme in patients with SLE and some of the drugs used in the treatment of SLE are among the other possible reasons for the higher prevalence of hyperuricemia in patients with SLE.

Studies have shown that increases in serum uric acid levels may be tied to an increased risk of cardiovascular disease and mortality. In addition, hyperuricemia has been shown to be associated with endothelial dysfunction as well as the oxidation of lipoproteins within atherosclerotic plaques (contributors to cardiovascular disease risk).

Several studies have highlighted the role of uric acid as an independent biomarker of cardiovascular disease risk. . The link between hyperuricemia and the risk of atherosclerotic cardiovascular and cerebrovascular disease has been well-established. .

In an observational cohort study testing the association between hyperuricemia and coronary artery calcification, the results showed that hyperuricemia is an independent risk factor for sub-clinical atherosclerosis in young adults .

Depending on the microenvironment, uric acid may act as an antioxidant or an oxidant. Under ischemic conditions, xanthine oxidase uses oxygen as an electron acceptor instead of nicotinamide adenine dinucleotide (NAD+) resulting in the formation of superoxide anion and hydrogen peroxide. Oxidants cause endothelial dysfunction by reacting with and removing nitric oxide (NO), which prevents vasodilation of the endothelium. This promotes a pro-inflammatory state that causes endothelial dysfunction and contributes to atherosclerosis and cardiovascular disease .Uric acid can also induce vascular smooth muscle cell proliferation in vitro by producing pro-inflammatory, pro-oxidative, and vasoconstrictive substances. Uric acid stimulates the production of monocyte chemoattractant protein-1 (MCP-1), a chemokine involved in atherosclerosis. Increased production of MCP-1 increases cell proliferation and production of pro-inflammatory mediators. Uric acid stimulates monocyte chemoattractant protein-1 production in vascular smooth muscle cells via mitogen-activated protein kinase and cyclooxygenase-2 .

This study aims to emphasize the role of flow mediated dilation in the detection of endothelial dysfunction in SLE patients and linking it to hyperuricemia as a predictor and contributor of cardiovascular affection which can be useful to guide therapeutic decisions in these patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* female patient with SLE aged more than 18

Exclusion Criteria:

* male patients
* patient with established cardiovascular disease, patients with end stage renal disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: femals patient whose age from 18 to 45yrs old
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2022-12-27 (Estimated); Study Completion 2023-12-27 (Estimated)

PRIMARY OUTCOMES:
percentage of SLE patients who have premature atherosclerosis based on abnormal flow mediated dilation FMD in assiciation with hyperuricemia as predictors of cardiovascular affection in SLE patient | about 1 yrs
percentage of hyperuricemic patients wh have premature atherosclerosis based on flow mediated dilation | about 1 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Rafaat fathy, Principal Investigator — Rafaatfathy@yahoo.com
Locations (1):
- Assuit University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hayden MR, Tyagi SC. Uric acid: A new look at an old risk marker for cardiovascular disease, metabolic syndrome, and type 2 diabetes mellitus: The urate redox shuttle. Nutr Metab (Lond). 2004 Oct 19;1(1):10. doi: 10.1186/1743-7075-1-10. PMID 15507132
- [Background] Crawley WT, Jungels CG, Stenmark KR, Fini MA. U-shaped association of uric acid to overall-cause mortality and its impact on clinical management of hyperuricemia. Redox Biol. 2022 May;51:102271. doi: 10.1016/j.redox.2022.102271. Epub 2022 Feb 17. PMID 35228125